CLINICAL TRIAL: NCT07183540
Title: Study on the Effect of Ultra-early Autologous Cranioplasty on Neurological Function Recovery: a Multicenter, Prospective, Open-label, Endpoint-blinded, Randomized Controlled Study
Brief Title: Study on the Effect of Ultra-early Autologous Cranioplasty on Neurological Function Recovery
Acronym: FAST-ECP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital Of Guizhou Medical University (Other)
Responsible Party: Principal Investigator, Kaya Xu, Principal Investigator, The Affiliated Hospital Of Guizhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YE2025NW-140
Record Dates: First submitted 2025-09-11; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Cranial Defect
Keywords: Decompressive craniectomy and Cranioplasty; operation opportunity; ultra-early; Autologous skull

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study was open-label, endpoint-blinded, i.e. only the patients themselves and the treating physicians knew the randomization assignment results, baseline was evaluated by investigators who did not know the actual patient assignment, and primary endpoint visits were conducted by trained third parties who did not know what treatment the patients received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The autologous skull repair surgery will be completed within 6 weeks after the DC operation.
  Interventions: Procedure: operation opportunity-within 6 weeks after the DC operation.
- control group (Active Comparator): The surgery should be completed within 90 to 180 days after DC.
  Interventions: Procedure: operation opportunity-within 90 to 180 days after the DC operation.

INTERVENTIONS:
Procedure: operation opportunity-within 6 weeks after the DC operation. — The autologous skull repair surgery will be completed within 6 weeks after the DC operation.
  Arms: experimental group
Procedure: operation opportunity-within 90 to 180 days after the DC operation. — The autologous skull repair surgery should be completed within 90 to 180 days after DC.
  Arms: control group

SUMMARY:
To compare the neurological recovery and complication rate of autogenous cranioplasty(CP) within 6 weeks after decompressive craniectomy (DC) with that of autogenous cranioplasty within 3~6 months after DC.

DETAILED DESCRIPTION:
Objective:

To compare the neurological recovery and complication rate of autogenous cranioplasty(CP) within 6 weeks after decompressive craniectomy (DC) with that of autogenous cranioplasty within 3~6 months after DC.

Design:

This study is a multi-center, prospective, randomized controlled, open-label trial.

Interventions:

Intervention measures were the time point of cranioplasty: within 6 weeks after decompressive craniectomy VS 3-6 months after decompressive craniectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Decompressive craniectomy due to craniocerebral trauma, cerebral ischemia and cerebral hemorrhage.
2. Age 18 - 80 years.
3. The first time for cranial repair.
4. unilateral skull defect.
5. Compliant with recommended decompressive bone flap surgery and autogenous decompressive bone flap after bone flap collection
6. signed the informed consent.

Exclusion Criteria:

1. Poor healing of skin flap (active infection, non-healing, necrosis, sinus, thin or poor blood supply, etc.).
2. Fracture of bone flap ≥2 pieces, partial open fracture
3. Intracranial infection before operation.
4. Severe bone metabolic diseases.
5. Long-term use of immunosuppressants.
6. Pregnant or lactating women.
7. Coagulation disorders.
8. Severe cardiopulmonary insufficiency.
9. It is estimated that the CP process cannot be completed within 6 weeks after the bone plate decompression surgery.
10. Skull defect size less than 25cm².
11. Life expectancy less than 1 year.
12. mRS greater than 1 before primary disease.
13. Diabetic patients.
14. Patients who are unable to cooperate with follow-up assessment (e.g. mental illness).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 582 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale (mRS) 0-2 | at 180 (± 7) days
  The proportion of patients with a modified Rankin Scale (mRS) score of ≤ 2

SECONDARY OUTCOMES:
mRS≤2 and mRS ≤3 | 90 (±7) days after CP
  Proportion of mRS≤2 and proportion of mRS ≤3
mRS ≤3 | 180 (±7) days after CP
  Proportion of mRS≤2 and proportion of mRS ≤3
Mini-Mental State Examination (MMSE) score | 90 days (±7 days) and 180 days (±7 days) after CP surgery
  Minimum score 0 and maximum score 30 with higher score being better outcome
Glasgow Outcome Score (GOS) | 90 days (±7 days) and 180 days (±7 days) after CP surgery
  Minimum score 1 and maximum score 8 with higher number being better outcome
hydrocephalus or Cerebrospinal fluid shunt surgery rate | 90 days (±7 days) and 180 days (±7 days) after CP surgery
  The incidence of hydrocephalus or CSF shunt surgery
Total medical expenses (excluding materials) | At the time of discharge from CP, 90 (±7) days after CP-CP and 180 (±7) days after CP-CP at discharge
Complications related medical expenses | At the time of discharge from CP, 90 (±7) days after CP-CP and 180 (±7) days after CP-CP at discharge
Incidence of infection, poor healing, and subcutaneous effusion | 90 days (±7 days) and 180 days (±7 days) after CP surgery
The incidence rate of intracranial hemorrhage | 90 days (±7 days) and 180 days (±7 days) after CP surgery
incidence of epilepsy | 90 days (±7 days) and 180 days (±7 days) after CP surgery
incidence of reoperation | 90 days (±7 days) and 180 days (±7 days) after CP surgery

OTHER OUTCOMES:
Overall mortality rate | 180 (±7) days after CP surgery
  All etiology of mortality

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Anshun People's Hospital (Ward One), Anshun, Guizhou
  - Anshun People's Hospital (Ward Two), Anshun, Guizhou
  - The First People's Hospital of Bijie City, Bijie, Guizhou
  - Guizhou Provincial Workers' Hospital, Guiyang, Guizhou
  - Qianfengdong Prefecture People's Hospital, Kaili, Guizhou
  - Zunyi Medical University Affiliated Hospital, Zunyi, Guizhou
  - Neijiang First People's Hospital, Neijiang, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morton RP, Abecassis IJ, Hanson JF, Barber JK, Chen M, Kelly CM, Nerva JD, Emerson SN, Ene CI, Levitt MR, Chowdhary MM, Ko AL, Chesnut RM. Timing of cranioplasty: a 10.75-year single-center analysis of 754 patients. J Neurosurg. 2018 Jun;128(6):1648-1652. doi: 10.3171/2016.11.JNS161917. Epub 2017 Aug 11. PMID 28799868
- [Background] Eaton JC, Greil ME, Nistal D, Caldwell DJ, Robinson E, Aljuboori Z, Temkin N, Bonow RH, Chesnut RM. Complications associated with early cranioplasty for patients with traumatic brain injury: a 25-year single-center analysis. J Neurosurg. 2022 Jan 21;137(3):776-781. doi: 10.3171/2021.11.JNS211557. Print 2022 Sep 1. PMID 35061995
- [Background] Mirabet V, Garcia D, Yague N, Larrea LR, Arbona C, Botella C. The storage of skull bone flaps for autologous cranioplasty: literature review. Cell Tissue Bank. 2021 Sep;22(3):355-367. doi: 10.1007/s10561-020-09897-2. Epub 2021 Jan 9. PMID 33423107
- [Background] Piedra MP, Ragel BT, Dogan A, Coppa ND, Delashaw JB. Timing of cranioplasty after decompressive craniectomy for ischemic or hemorrhagic stroke. J Neurosurg. 2013 Jan;118(1):109-14. doi: 10.3171/2012.10.JNS121037. Epub 2012 Nov 9. PMID 23140156
- [Background] Malcolm JG, Rindler RS, Chu JK, Chokshi F, Grossberg JA, Pradilla G, Ahmad FU. Early Cranioplasty is Associated with Greater Neurological Improvement: A Systematic Review and Meta-Analysis. Neurosurgery. 2018 Mar 1;82(3):278-288. doi: 10.1093/neuros/nyx182. PMID 28419358
- [Background] Huang YH, Lee TC, Yang KY, Liao CC. Is timing of cranioplasty following posttraumatic craniectomy related to neurological outcome? Int J Surg. 2013;11(9):886-90. doi: 10.1016/j.ijsu.2013.07.013. Epub 2013 Aug 7. PMID 23933129
- [Background] Yamada A, Imai K, Nomachi T, Fujimoto T, Sakamoto H, Kitano S. Cranial distraction for plagiocephaly: quantitative morphologic analyses of cranium using three-dimensional computed tomography and a life-size model. J Craniofac Surg. 2005 Jul;16(4):688-93. doi: 10.1097/01.scs.0000168995.27882.66. PMID 16077318
- [Background] Hokugo A, Sawada Y, Sugimoto K, Fukuda A, Mushimoto K, Morita S, Tabata Y. Preparation of prefabricated vascularized bone graft with neoangiogenesis by combination of autologous tissue and biodegradable materials. Int J Oral Maxillofac Surg. 2006 Nov;35(11):1034-40. doi: 10.1016/j.ijom.2006.06.003. Epub 2006 Sep 11. PMID 16965895
- [Background] Martin MP, Olson S. Post-operative complications with titanium mesh. J Clin Neurosci. 2009 Aug;16(8):1080-1. doi: 10.1016/j.jocn.2008.07.087. Epub 2009 May 7. PMID 19427221
- [Background] Gooch MR, Gin GE, Kenning TJ, German JW. Complications of cranioplasty following decompressive craniectomy: analysis of 62 cases. Neurosurg Focus. 2009 Jun;26(6):E9. doi: 10.3171/2009.3.FOCUS0962. PMID 19485722
- [Background] Taub PJ, Rudkin GH, Clearihue WJ 3rd, Miller TA. Prefabricated alloplastic implants for cranial defects. Plast Reconstr Surg. 2003 Mar;111(3):1233-40. doi: 10.1097/01.PRS.0000046048.77472.23. No abstract available. PMID 12621197
- [Background] Lilja-Cyron A, Andresen M, Kelsen J, Andreasen TH, Fugleholm K, Juhler M. Long-Term Effect of Decompressive Craniectomy on Intracranial Pressure and Possible Implications for Intracranial Fluid Movements. Neurosurgery. 2020 Feb 1;86(2):231-240. doi: 10.1093/neuros/nyz049. PMID 30768137
- [Background] Winkler PA, Stummer W, Linke R, Krishnan KG, Tatsch K. Influence of cranioplasty on postural blood flow regulation, cerebrovascular reserve capacity, and cerebral glucose metabolism. J Neurosurg. 2000 Jul;93(1):53-61. doi: 10.3171/jns.2000.93.1.0053. PMID 10883905
- [Background] Kuo JR, Wang CC, Chio CC, Cheng TJ. Neurological improvement after cranioplasty - analysis by transcranial doppler ultrasonography. J Clin Neurosci. 2004 Jun;11(5):486-9. doi: 10.1016/j.jocn.2003.06.005. PMID 15177389
- [Background] Yamaura A, Makino H. Neurological deficits in the presence of the sinking skin flap following decompressive craniectomy. Neurol Med Chir (Tokyo). 1977;17(1 Pt 1):43-53. doi: 10.2176/nmc.17pt1.43. No abstract available. PMID 74031
- [Background] Hutchinson PJ, Kolias AG, Timofeev IS, Corteen EA, Czosnyka M, Timothy J, Anderson I, Bulters DO, Belli A, Eynon CA, Wadley J, Mendelow AD, Mitchell PM, Wilson MH, Critchley G, Sahuquillo J, Unterberg A, Servadei F, Teasdale GM, Pickard JD, Menon DK, Murray GD, Kirkpatrick PJ; RESCUEicp Trial Collaborators. Trial of Decompressive Craniectomy for Traumatic Intracranial Hypertension. N Engl J Med. 2016 Sep 22;375(12):1119-30. doi: 10.1056/NEJMoa1605215. Epub 2016 Sep 7. PMID 27602507